CLINICAL TRIAL: NCT00335205
Title: A Placebo Controlled Trial of the Dopamine D-2 Receptor Agonist Ropinirole in Treatment of 60 Patients With Refractory Bipolar I and II Depression.
Brief Title: A Placebo Controlled Trial of the Dopamine D-2 Receptor Agonist Ropinirole in Treatment of 60 Patients With Refractory Bipolar Depression.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Jerusalem Mental Health Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-02-2690-LG-CTIL
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2006-06

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: ropinirole; dopamine; D2; depression; bipolar
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Depression | interventions — ropinirole

INTERVENTIONS:
Drug: ropinirole

SUMMARY:
We hypothesize that depressed patients who have not responded to their current antidepressant medication will respond to the addition of ropinirole to their current regimen at a rate better than placebo.

DETAILED DESCRIPTION:
Most pharmacologic treatments of depression rely on serotonergic and/or noradrenergic mechanisms. Yet, evidence both from animal studies and from human trials suggests a role for dopaminergic pathways and particularly for dopamine D2-like receptors in the treatment of depression. In recent years, two new selective agonists of dopamine D2-like receptors have come into clinical use for the treatment of parkinsonism. Preliminary evidence suggests that these drugs might be useful as antidepressants. We are testing whether one of these agonists, ropinirole, is an effective augmentation strategy in depressed patients in a double-blind, randomized, controlled trial. We are recruiting unipolar and bipolar patients who remained depressed (modified Hamilton Depression Rating Scale score greater than 16) despite at least 4 weeks of treatment with an adequate dose of antidepressant medication. Patients receive either 2mg of oral ropinirole or placebo twice daily added on to their current medication and are evaluated weekly over 7 weeks and are assessed weekly using two depression rating scales.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depression OR Bipolar I or II Disorder - Currently Depressed
* One month of a stable, adequate dose of antidepressant medication
* Bipolar patients must have a mood stabilizer
* At least 18 years old
* Modified HDRS-21 more than 16 (Scores reverse vegetative symptoms.)
* Informed Consent

Exclusion Criteria:

* CVA
* Antipsychotic Medication
* Drug or Alcohol Abuse
* Active Suicidality
* Rapid Cycling Bipolar Disorder
* Neurologic or Dementing Illness
* Psychosis
* Parkinsonism
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale Score

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale Score

CONTACTS AND LOCATIONS:
Overall Officials: Leon Grunhaus, MD, Principal Investigator — Jerusalem Mental Health Center
Locations (2):
- Israel (2):
  - Jerusalem Mental Health Center, Jerusalem
  - Chaim Sheba Medical Center, Dept. of Psychiatry, Tel Litwinsky